CLINICAL TRIAL: NCT05799742
Title: Bilateral Inguinal Hernia Repair and Male Fertility: A Randomized Clinical Trial Comparing Lichtenstein Versus Laparoscopic Transabdominal Preperitoneal (TAPP) Technique
Brief Title: Inguinal Hernia Repair and Male Fertility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 45535015.40000.0068
Record Dates: First submitted 2023-02-17; First posted 2023-04-05 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2019-01

CONDITIONS: Inguinal Hernia Bilateral
Keywords: Inguinal hernia; Infertility; Laparoscopy
MeSH Terms: conditions — Hernia, Inguinal; Infertility

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial with two groups, in according to hernioplasty correction approach
Who Masked: Outcomes Assessor
Masking Description: Masking couldn't be possible because of the surgical technique
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lichtenstein (Active Comparator): Conventional approach
  Interventions: Procedure: Bilateral hernioplasty
- Laparoscopy (Experimental): Experimental approach
  Interventions: Procedure: Bilateral hernioplasty

INTERVENTIONS:
Procedure: Bilateral hernioplasty

SUMMARY:
General objective: To evaluate the fertility of adult men submitted to bilateral herniorrhaphy with mesh placement by the Lichtenstein and laparoscopic approaches

DETAILED DESCRIPTION:
Specific objectives: To correlate pre and postoperative data (90 and 180 days) of adult men, according to biochemistry parameters (hemogram and CRP), autoimmune (anti-sperm antibodies), hormonal (FSH, LH and testosterone), perfusion and volume testicular (USG of testicles with Doppler), spermogram, sexual changes, pain and quality of life (standard questionnaires).

ELIGIBILITY:
Inclusion Criteria:

* Male
* Age between 19 and 60 years old
* Bilateral inguinal hernia
* Primary and reducible inguinal hernia

Exclusion Criteria:

* Age less than 19 or more than 60 years old
* ASA >III
* Genito-urinary infection
* Immunodeficiency
* History of testicular trauma2
* History of surgery or pelvic radiotherapy
* History of testicular disease
* Fertility problems or sexual
* Illness that can be infertile
* Recurrent hernia
* Unilateral hernia
* Femoral or inguine-scrotal hernia
* Imprisoned hernia
* Use of Gonadotrophins
* Use of anabolic steroids

Ages: 19 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-12-15 (Actual)

PRIMARY OUTCOMES:
Sperm Volume | Preoperative
  Sperm Volume (in ml) measured by Semen analysis
Sperm concentration | Preoperative
  Sperm concentration (million sperm/ml) measured by Semen analysis
Sperm number | Preoperative
  Sperm number in million measured by Semen analysis
Sperm motility | Preoperative
  Sperm motility in % of progression measured by Semen analysis
Sperm morphology | Preoperative
  Sperm morphology, according to the Kruger classification, evaluated by Semen analysis
Testicular volume | Preoperative
  Testicular volume, in cm3, measured by testicular ultrasound
Testicular vascularization | Preoperative
  Testicular vascularization, normal or not, measured by testicular Doppler ultrasound
Sperm Volume | 90th postoperative day
  Sperm Volume (in ml) measured by Semen analysis
Sperm concentration | 90th postoperative day
  Sperm concentration (million sperm/ml) measured by Semen analysis
Sperm number | 90th postoperative day
  Sperm number in million measured by Semen analysis
Sperm motility | 90th postoperative day
  Sperm motility in % of progression measured by Semen analysis
Sperm morphology | 90th postoperative day
  Sperm morphology, according to the Kruger classification, evaluated by Semen analysis
Testicular volume | 90th postoperative day
  Testicular volume, in cm3, measured by testicular ultrasound
Testicular vascularization | 90th postoperative day
  Testicular vascularization, normal or not, measured by testicular Doppler ultrasound
Sperm Volume | 180th postoperative day
  Sperm Volume (in ml) measured by Semen analysis
Sperm concentration | 180th postoperative day
  Sperm concentration (million sperm/ml) measured by Semen analysis
Sperm number | 180th postoperative day
  Sperm number in million measured by Semen analysis
Sperm motility | 180th postoperative day
  Sperm motility in % of progression measured by Semen analysis
Sperm morphology | 180th postoperative day
  Sperm morphology, according to the Kruger classification, evaluated by Semen analysis
Semen analysis | 180th postoperative day
  Volume (ml), Concentration (million/ml), Sperm number (million), Motility (% of progression), Morphology (Kruger classification)
Testicular volume | 180th postoperative day
  Testicular volume, in cm3, measured by testicular ultrasound
Testicular vascularization | 180th postoperative day
  Testicular vascularization, normal or not, measured by testicular Doppler ultrasound

SECONDARY OUTCOMES:
Follicle Stimulating Hormone (FSH) dosage | Preoperative
  Serum FSH (IU/L)
Luteinizing Hormone (LH) dosage | Preoperative
  Serum LH (IU/L)
Testosterone Hormone dosage | Preoperative
  Serum Testosterone (ng/dl)
Sex hormone-binding globulin (SHGB) dosage | Preoperative
  Serum SHGB (nmol/L)
Sexual activity | Preoperative
  Satisfied or not with sexual performance, Changes in arousal, Changes in libido and Changes in ejaculation or orgasm (Specific questionnaires)
Quality-of-life evaluation (SF-36 questionnaire) | Preoperative
  SF36 Domains: Role physical, Physical function, Role emotional, Energy, Emotional health, Social functioning, Bodily pain and General health. Scale ranging from 0 to 100, where zero is the worst state and 100 is the best.
Postoperative pain | 7th postoperative day
  Visual Analog Scale (VAS) score ranging from 0 to 10, with 0 indicating no pain and 10 indicating the worst possible pain
Postoperative pain | 30th postoperative day
  Visual Analog Scale (VAS) score ranging from 0 to 10, with 0 indicating no pain and 10 indicating the worst possible pain
Follicle Stimulating Hormone (FSH) dosage | 90th postoperative day
  Serum FSH (IU/L)
Luteinizing Hormone (LH) dosage | 90th postoperative day
  Serum LH (IU/L)
Testosterone Hormone dosage | 90th postoperative day
  Testosterone (ng/dl)
Sex hormone-binding globulin (SHGB) dosage | 90th postoperative day
  Serum SHGB (nmol/L)
Sexual activity | 90th postoperative day
  Satisfied or not with sexual performance, Changes in arousal, Changes in libido and Changes in ejaculation or orgasm (Specific questionnaires)
Quality-of-life evaluation (SF-36 questionnaire) | 90th postoperative day
  SF36 Domains: Role physical, Physical function, Role emotional, Energy, Emotional health, Social functioning, Bodily pain and General health. Scale ranging from 0 to 100, where zero is the worst state and 100 is the best.
Postoperative pain | 90th postoperative day
  Visual Analog Scale (VAS) score ranging from 0 to 10, with 0 indicating no pain and 10 indicating the worst possible pain
Follicle Stimulating Hormone (FSH) dosage | 180th postoperative day
  Serum FSH (IU/L)
Luteinizing Hormone (LH) dosage | 180th postoperative day
  Serum LH (IU/L)
Testosterone Hormone dosage | 180th postoperative day
  Serum Testosterone (ng/dl)
Sex hormone-binding globulin (SHGB) dosage | 180th postoperative day
  Serum SHGB (nmol/L)
Sexual activity | 180th postoperative day
  Satisfied or not with sexual performance, Changes in arousal, Changes in libido and Changes in ejaculation or orgasm (Specific questionnaires)
Quality-of-life evaluation (SF-36 questionnaire) | 180th postoperative day
  SF36 Domains: Role physical, Physical function, Role emotional, Energy, Emotional health, Social functioning, Bodily pain and General health. Scale ranging from 0 to 100, where zero is the worst state and 100 is the best.
Postoperative pain | 180th postoperative day
  Visual Analog Scale (VAS) score ranging from 0 to 10, with 0 indicating no pain and 10 indicating the worst possible pain

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data that underlie individual participant data that underlie collected during the trial, after deidentification (text, tables, figures, and appendices) will be shared. Study Protocol also will be available. Data will be available immediately following publication, no end dates, to anyone who wishes to access the data, for any types of analyses. Proposals should be directed to sergio.damous@hc.fm.usp.br
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available immediately following publication, no end dates.
Access Criteria: Proposals should be directed to sergio.damous@hc.fm.usp.br

REFERENCES:
- [Derived] Damous SHB, Damous LL, Borges VA, Fontella AK, Miranda JDS, Koike MK, Saito OC, Birolini CAV, Utiyama EM. Bilateral inguinal hernia repair and male fertility: a randomized clinical trial comparing Lichtenstein versus laparoscopic transabdominal preperitoneal (TAPP) technique. Surg Endosc. 2023 Dec;37(12):9263-9274. doi: 10.1007/s00464-023-10499-8. Epub 2023 Oct 25. PMID 37880447